CLINICAL TRIAL: NCT05462691
Title: "It is Necessary to Suture the Tuberosities in Inverted Prostheses Implanted for Acute Fractures of the Proximal Humerus?. Prospective Randomized Study
Brief Title: "Suture of the Tuberosities in Inverted Prostheses" Implanted for Acute Fractures of the Proximal Humerus?.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Clinical Professor, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/10519
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Proximal Humeral Fractures, Reverse Shoulder Prostheses, Tuberosities
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: prospective randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: patients will be blinded to the assignment group. outcomes assessors will be blinded to the assignment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without tuberosity reconstruction (Experimental): patients undergoing reverse shoulder arthroplasty because a proximal humeral fracture with suturing of the tuberosities
  Interventions: Procedure: tuberosity suture
- Patients with tuberosity reconstruction (Active Comparator): patients undergoing reverse shoulder arthroplasty because a proximal humeral fracture without suturing of the tuberosities
  Interventions: Procedure: tuberosity suture

INTERVENTIONS:
Procedure: tuberosity suture — to suture or not suture the tuberosities in reverse shoulder arthroplasty because of a proximal humeral fracture

SUMMARY:
Complex fractures of the proximal humerus in elderly patients constitute a growing problem. Osteoporosis linked to these fractures prevents osteosynthesis correctly, so that if the offset between the fragments is large, it is necessary to implant a prosthesis. Inverted prostheses, normally used for the treatment of osteoarthritis with absence of the rotator cuff, have become the treatment of choice in these fractures obtaining very favorable results. Traditionally, once the prosthesis is implanted, they are sutured the tuberosities with the rotator cuff tendons to the prosthesis. This gesture is supposed to will improve patient function. However, this prosthesis was originally designed for use in patients without a rotator cuff, so the need for this suture, which lengthens surgical time and requires an increase in the number of sutures, which can potentially increase the risk of infection. With the results of this study, it would be possible to reduce the surgical time, the number of inert materials implanted, and potentially the risk of infection.

DETAILED DESCRIPTION:
Complex fractures of the proximal humerus in elderly patients constitute a growing problem. Osteoporosis linked to these fractures prevents osteosynthesis correctly, so that if the offset between the fragments is large, it is necessary to implant a prosthesis. Inverted prostheses, normally used for the treatment of osteoarthritis with absence of the rotator cuff, have become the treatment of choice in these fractures obtaining very favorable results. Traditionally, once the prosthesis is implanted, they are sutured the tuberosities with the rotator cuff tendons to the prosthesis. This gesture is supposed to will improve patient function. However, this prosthesis was originally designed for use in patients without a rotator cuff, so the need for this suture, which lengthens surgical time and requires an increase in the number of sutures, which can potentially increase the risk of infection. With the results of this study, it would be possible to reduce the surgical time, the number of inert materials implanted, and potentially the risk of infection.

Primary objective:

To determine if there are differences in the perception of quality of life measured by through the Simple Shoulder Test scale, among the patients in whom sutured the tuberosities and patients who have had the tuberosities excised tuberosities.

Secondary objectives:

To determine if there are differences between the patients in whom suturing has been the tuberosities and patients who have had their tuberosities excised about:

* SPADI quality of life test.
* Constant functional test.
* number of prosthetic dislocations
* Percentage of scapular notch development measured according to the Sirveaux scale.
* Number of dislocations.
* number of infections.
* number of revision surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients > 65 yrs. and < 85 yrs.
* Acute fracture of the proximal humerus.
* implantation of inverted shoulder prosthesis.

Exclusion Criteria:

* acute fractures of more than 3 weeks of evolution
* Associated fractures.
* senile dementia and/or cognitive alterations that prevent compliance protocols

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Simple Shoulder Test | 24 months
  Primary objective:
  To determine if there are differences in the perception of quality of life measured by through the Simple Shoulder Test scale, among the patients in whom sutured the tuberosities and patients who have had the tuberosities excised tuberosities.

IPD SHARING:
Plan to Share IPD: Undecided